CLINICAL TRIAL: NCT03415139
Title: Islet Cell and ST2 Axis Dysregulation in Post-Transplant Diabetes Mellitus
Brief Title: Finding the Cause for Post-Transplant Diabetes Mellitus After Allogeneic Hematopoietic Cell Transplant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Brian Engelhardt, MD, Associate Professor of Medicine, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC CTT 1836
Record Dates: First submitted 2018-01-15; First posted 2018-01-30 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus; Cancer
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum / plasma and peripheral blood mononuclear cells will be collected before and after hematopoietic stem cell transplant (HCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1 for MRD HCT Recipients: Patients undergo an Oral Glucose Tolerance Test (OGTT) and 1 hyperglycemic clamp will be performed on separate days prior to transplant and then each procedure will be repeated once between day+80 to day+100 (+/- 10 days) after transplant.
  Interventions: Drug: Oral Glucose Tolerance Test (OGTT); Drug: Hyperglycemic clamp procedure
- Arm 2 for MRD HCT Recipients: Patients undergo 2 Oral Glucose Tolerance Test (OGTTs) (with and without GLP-1 analogue) will be performed on separate days prior to transplant and then each procedure will be repeated once between day+80 to day+100 (+/- 10 days) after transplant.
  Interventions: Drug: 2 OGTTs with and without GLP-1 analogue

INTERVENTIONS:
Drug: Oral Glucose Tolerance Test (OGTT) — A standard OGTT will be performed. During OGTT 75gm of glucose will be given followed by phlebotomy.
  Groups: Arm 1 for MRD HCT Recipients
Drug: 2 OGTTs with and without GLP-1 analogue — A standard OGTT will be performed and a second OGTT procedure will be repeated on a different day with GLP-1 analogue.
  Groups: Arm 2 for MRD HCT Recipients
Drug: Hyperglycemic clamp procedure — During the hyperglycemic clamp procedure, D20 will given, followed by phlebotomy.
  Groups: Arm 1 for MRD HCT Recipients

SUMMARY:
This clinical research studies the physiology and immunology of new-onset post-transplant diabetes mellitus in patients undergoing allogeneic stem cell transplantation. Oral glucose tolerance tests (OGTT), hyperglycemic clamps, and immune assays will be used to define the mechanisms associated with abnormal glucose homeostasis following stem cell transplantation. Information from this clinical trial could be used to develop standardized screening procedures or to develop optimal treatment strategies for patients developing post-transplant diabetes mellitus.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if changes in islet cell physiology are detectable before or after matched related donor (MRD) hematopoietic stem cell transplant (HCT) in patients developing new-onset post-transplant diabetes mellitus (PTDM).

1. To determine if a compensatory increase in glucose stimulated insulin secretion (GSIS) by β-cells precedes PTDM development in patients without diabetes undergoing MRD HCT.
2. To determine if excess glucagon secretion and impaired α-cell response to glucose or GLP-1 contributes to the hyperglycemia of PTDM.

II. To determine if the IL-33/ST2 axis promotes immune/islet cell dysregulation during PTDM.

OUTLINE:

Patients undergo 2 OGTTs and a standard hyperglycemic clamp procedure prior to HCT. Patients then undergo repeat OGTTs and a hyperglycemic clamp procedure once after HCT between days 80-100.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Patients undergoing allogeneic hematopoietic stem cell transplantation (HCT).

Exclusion Criteria for Patients:

* Patients who have not received an allogeneic HCT
* Recent or current history of diabetes mellitus, defined as:1) diabetes therapy within 6 months of enrollment, or 2) fasting blood glucose at "pre-admit" (screening) visit >= 126 mg/dL
* Pregnancy or breastfeeding
* Umbilical cord blood transplants
* Patients on established, chronic corticosteroid therapy (> 10 mg /day of prednisone or prednisone equivalent) prior to transplant; established, chronic corticosteroid therapy is defined as daily dosing of > 10 mg/day of prednisone or prednisone equivalent for at least 2 weeks prior to the start of conditioning/chemotherapy or plans to continue pre-transplant corticosteroids (> 10 mg/day of prednisone or prednisone equivalent) indefinitely after transplantation
* Inability to give informed consent
* Any condition which, in the opinion of the investigator, might interfere with study objective
* Any reason which, in the opinion of the investigator, adds additional risk to the patient

Additional exclusion criteria (Arms 1 and 2 Aim 1 only):

-Diagnosis of diabetes by standard oral glucose tolerance testing prior to transplant (2-hour plasma glucose value ≥ 200 mg/dL) in either Arm 1 or 2 will exclude further testing as per Aim 1. Immunological / metabolic testing as per Aim 2 will still be allowed

DONORS Inclusion Criteria for Donors (Arm 1 and Arm 2) Donors undergoing stem cell collection for related allogeneic stem cell transplant

Exclusion Criteria for Donors (Arms 1 and 2):

* Individuals not donating stem cells
* Pregnancy or breastfeeding
* Inability to give informed consent
* Any condition which, in the opinion of the investigator, might interfere with study objective

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without a history of diabetes mellitus undergoing allogeneic hematopoietic stem cell transplantation (HCT).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Pre-transplant insulin secretion will be measured as glucose stimulated insulin secretion (GSIS) during a hyperglycemic clamp procedure among patients who do or do not go on to develop PTDM (univariable analysis). | Up to 28 days pre-transplant
  A hyperglycemic clamp procedure will be performed pre-transplant. Pre-transplant will be defined as no more than 28 days before allogeneic hematopoietic cell transplantation. Patients will then be followed for 100 days after transplant for development of diabetes. In univariable analysis, a Wilcoxon rank sum test will be applied to compare the population mean difference in GSIS between these two groups.
Pre-transplant insulin secretion will be measured as glucose stimulated insulin secretion (GSIS) during a hyperglycemic clamp procedure among patients who do or do not go on to develop PTDM (multivariable analysis). | Up to 28 days pre-transplant
  A hyperglycemic clamp procedure will be performed pre-transplant. Pre-transplant will be defined as no more than 28 days before allogeneic hematopoietic cell transplantation. Patients will then be followed for 100 days after transplant for development of diabetes. In multivariable analysis, logistic regression will evaluate whether GSIS is an independent predictor of PTDM after adjusting for the following covariates: gender, conditioning (ablative vs. reduced intensity), or acute graft-versus-host disease (GVHD) requiring steroids. The estimated odds ratio (OR) and 95% confidence interval of the OR will be provided to measure the effect of the association.
Post-transplant glucagon secretion will be measured during the oral glucose tolerance test among patients who do or do not develop PTDM (univariable analysis). | Up to 100 days after transplant
  Patients will be followed for 100 days after transplant for development of diabetes. In univariable analysis, a Wilcoxon rank sum test will be applied to compare the population mean difference in glucagon secretion between these two groups.
Post-transplant glucagon secretion will be measured during the oral glucose tolerance test among patients who do or do not develop PTDM (multivariable analysis). | Up to 100 days after transplant
  Patients will be followed for 100 days after transplant for development of diabetes. In multivariable analysis, a logistic regression will evaluate whether glucagon secretion is independently associated with PTDM after adjusting for the following covariates: gender, conditioning (ablative vs. reduced intensity), or acute graft-versus-host disease (GVHD) requiring steroids. The estimated odds ratio (OR) and 95% confidence interval of the OR will be provided to measure the effect of the association.
Plasma IL-33 levels will be measured among patients who do or do not develop PTDM (univariable analysis). | Up to 100 days after transplant
  Patients will be followed for 100 days after transplant for development of diabetes. In univariable analysis, a Wilcoxon rank sum test will be applied to compare the population mean difference in IL-33 between these two groups.
Plasma IL-33 levels will be measured among patients who do or do not develop PTDM (multivariable analysis). | Up to 100 days after transplant
  In multivariable analysis, logistic regression will evaluate whether IL-33 is independently associated with PTDM after adjusting for the following covariates: gender, conditioning (ablative vs. reduced intensity), or acute graft-versus-host disease (GVHD) requiring steroids. The estimated odds ratio (OR) and 95% confidence interval of the OR will be provided to measure the effect of the association.

CONTACTS AND LOCATIONS:
Overall Officials: Brian G. Engelhardt, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03415139/Prot_SAP_000.pdf